CLINICAL TRIAL: NCT04801030
Title: Using Multi-strategies to Address COVID-19 Vaccine Hesitancy Among African Americans
Brief Title: COVID-19 Vaccine Hesitancy Among African Americans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meharry Medical College (Other)
Collaborators: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-03-1076
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Vaccine Refusal; Communication
MeSH Terms: conditions — COVID-19; Vaccination Refusal; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Culturally-appropriate social marketing campaign (Experimental): Participants will receive a multi-layered, social marketing campaign which is deemed culturally appropriate. This will occur over a 6 month -time period. Rates will be observed at 0, 6, and 12 months.
  Interventions: Behavioral: YourCoViDVaxFacts
- Control Arm 1 (No Intervention): Participants will receive no intervention, only to serve as a control site. Rates will be observed at 0, 6, and 12 months.
- Control Arm 2 (No Intervention): Participants will receive no intervention, only to serve as a control site. Rates will be observed at 0, 6, and 12 months.

INTERVENTIONS:
Behavioral: YourCoViDVaxFacts — The intervention will be delivered via multiple strategies- social media (YouTube, Facebook), radio, newspaper, tv ads, community partner networks. Participants receive culturally-tailored message on COVID-19 and the vaccine. The strategies will have a link that will open to a website that is optimized for viewing on a computer or mobile phone which has the look and feel of an app, but without requiring the user to download anything to the phone. On the website, participants will be prompted to select their top concerns from a list. Based on the responses, the top barriers or need will each be mapped to a corresponding educational message, which will be displayed to the user with appropriate images or graphics.
  Arms: Culturally-appropriate social marketing campaign

SUMMARY:
Coronavirus disease 2019 (COVID-19) has created a "state of emergency" for African Americans in the US. Recent findings indicate 31% of adults self-reported "wait and see" of the COVID-19 vaccine, of which 16% were African American. This project seeks to test the feasibility and impact of a multi-layered, culturally-appropriate social marketing intervention targeting COVID-19 vaccine hesitant (VH) African Americans to increase vaccine confidence, uptake, and completion of multi-dose vaccine series in Nashville/Davidson County, Tennessee. This study's novelty lies in being the first to assess feasibility and preliminary efficacy of a multi-layered, culturally-appropriate social marketing intervention to promote COVID-19 vaccination among African Americans in TN. Clinical significance is increased vaccine uptake and decreased COVID-19 burden and disparities.

DETAILED DESCRIPTION:
The goal of this application is to develop and test the feasibility and impact of a multi-layered, culturally-appropriate social marketing intervention targeting COVID-19 VH African Americans to increase uptake and completion of vaccine series in Nashville/Davidson County, Tennessee (TN). Investigators will partner with members of National Association for the Advancement of Colored People, Nashville Health Disparities Coalition, and Congregational Health Education Network to serve as an advisory committee. Investigators will also partner with Meharry Medical College (MMC) clinics and Tennessee Department of Health's (TDH) Immunization Program.

Aim 1. Engage with key stakeholders to develop a multi-layered, culturally-appropriate social marketing intervention targeting African Americans who are COVID-19 VH. Investigators will adapt an existing message library using the Health Belief Model,Theory of Reasoned Action, previous VH research, preliminary data of investigators, and feedback from community partners. Next, investigators will conduct semi-structured interviews with 25-30 VH individuals and 5-10 COVID-19 experts to elicit feedback on draft content. Qualitative data will be collected and analyzed iteratively, informing successive intervention modifications to cover a range of concerns for VH individuals, enhance message relevance, and determine media outlets for dissemination. Next, investigators will pre-test intervention prototypes with 16 COVID-19 VH individuals to make final modifications.

Aim 2a. Conduct a pilot study of the intervention and study protocol to demonstrate feasibility and assess impact. Investigators will conduct a pilot study using an experimental field trial design in three TN counties: Davidson County (1 intervention site) and Shelby and Hamilton Counties (2 control sites). COVID-19 vaccine uptake, primary outcome, assessed using: 1) aggregate data from partner clinics and TN immunization registry (TennIIS) and 2) individual, pre-post data from a marketing firm using random digit dialing (RDD). H1: COVID-19 vaccination rates will be higher for VH African Americans at intervention site compared to control sites. Implementation outcomes are feasibility, fidelity, acceptability, appropriateness, and penetration.

Aim 2b. To retrospectively explore knowledge, attitudes, intentions, and implementation outcomes post-intervention. Investigators will use qualitative methods to identify perceived acceptance of different types of media and webpage along with perceived change in knowledge, attitudes, and intentions from African Americans by degree of VH. Investigators will also explore appropriateness, feasibility, penetration, and fidelity as it relates to the social marketing intervention from 3 providers, 3 community-based organization (CBO) staff, and 2 TDH staff. Participants will be identified using RDD and community partner networks.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Unvaccinated for COVID-19
* Vaccine hesitant
* 18 years and older
* Speaks English

Exclusion Criteria:

* Not African American
* Receipt of COVID-19 vaccination
* under 18 years of age
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 6 months
  percent enrolled in study
Retention rates | 1 year
  percent completed baseline survey, percent completed follow-up survey
data collection processes | 1 year
  percent ascertained COVID 19 vaccine status post-intervention

SECONDARY OUTCOMES:
COVID-19 vaccine rates | 6 months
  Number of individuals vaccinated post-intervention
Attitudes toward COVID-19 vaccine | 6 months
  Change in attitudes toward COVID-19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Erves, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No